CLINICAL TRIAL: NCT05496946
Title: The Efficiency of Two Different Simulation Methods on Developing Head Bath Skills in Nursing Students
Brief Title: The Efficiency of Two Different Simulation Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Furkan Keles, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IMU16
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Nursing Education
Keywords: Nurse-Patient Relations; simulation; standardized patient

STUDY DESIGN:
Intervention Model Description: The sample size of the study; Using the G* Power 3.1.9.2 program, the mean and standard deviation of a similar study in the literature (İlaslan, 2019) (Spielberger State Anxiety Scale total score mean=28.8; SD=5.4 and Spielberger State Anxiety Scale total score mean=39, 5; SD=10.4). For the calculated effect size=0.91, α=0.05 and power=0.95, it was determined that there should be at least 33 students in both groups, for a total of 66 students. Students in the sample group were randomly assigned by the researcher to the Low-Reality Model (Experimental-1 Group) and Standardized Patient (Experimental-2 Group) groups.
Who Masked: Investigator
Masking Description: For randomization, a randomization table was created using the http://stattrek.com/statistics/random-numbergenerator.aspx site. As a result, the sample of the research; The purpose of the study was explained, and after the briefing, a total of 80 students, 40 students in both groups, who were allowed to participate in the research and who met the criteria for inclusion in the sample, formed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model with low proximity to reality group (Experimental): The students included in the experimental group 1 practiced the head bathing skill on a model with low proximity to reality. The model used here is a human model belonging to the Gaumard Scientific company with low proximity to reality.
  Interventions: Other: Head bathing skill
- Standardized patient Group (Experimental): The students in the experimental group 2 practiced the head bath skill on the standardized patient. A standardized patient is a healthy individual pretending to be a patient.
  Interventions: Other: Head bathing skill

INTERVENTIONS:
Other: Head bathing skill — A group of students will practice the head bathing skill in a model with low proximity to reality, while the students in the other group will practice on a healthy individual (Standardized patient) pretending to be patient.

SUMMARY:
In the literature, it is emphasized that the use of simulation improves the communication skills of the participants and that teamwork is important in providing patient safety and effective care. It is stated that students experience fear and anxiety in practice due to their lack of knowledge and clinical experience. Continuous repetitions and regular feedback provided by the trainings made by applying simulation increase the performance and self-confidence of the student. It is stated that the possibility of repeated application reduces the anxiety of the students. It is seen that different simulation types are used in the development of skills in nursing students in studies on this subject. As a result; It is seen that simulation has unlimited potential as an educational method and tool in nursing education. However; No study was found on a specific nursing practice and within the simulation scenario. of the study; In this study, it is aimed to evaluate the effectiveness of using standardized/simulated patient and low-fidelity patient models in head bath practice, which is one of the basic skills of nursing students. As a result of this study, the effective training method in the teaching of the head bath skill, which is taught within the scope of the nursing principles course, will be determined. In addition, it is thought that the periodical follow-up of the students (right after the teaching and at the end of the semester) and the permanence level of this education include a different aspect from other studies.

DETAILED DESCRIPTION:
There are different definitions in the literature about simulation. Gaba (2004) defines the simulation technique as "reminding or imitating important aspects of the real environment in an interactive way, accompanied by guides, in order to change or improve real experiences". Although there is no single definition of simulation, in general, simulation is a learning method in which a realistic model of an event or process is developed or imitated. Simulation in nursing education is a learning method applied in different ways to minimize the risks that students may encounter in the clinical setting.

There are many different types of simulations that provide knowledge and skills to nursing students, guide about the problems that may be encountered in the clinical environment, and are suitable for real situations. These are divided into low-tech simulation models, standard/simulated patient, computer-assisted simulations, virtual reality and touch systems, and integrated simulations.

The use of simulation in the nursing education curriculum has many advantages. The use of simulation in nursing education; By providing experience-based learning opportunities, it enables students to increase their self-confidence and improve their clinical decision-making skills. Students gain the ability to perform complete care, decision making, assessment, teamwork, skill development and management in a safe environment without misunderstanding the patient's current situation or fear of failure.

The use of simulation in nursing education is gaining importance in Turkey due to the increase in the number of students, insufficient clinical areas and ensuring patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year student of a nursing undergraduate program,
* To be taking the Nursing Basic Principles and Practices course for the first time,
* Getting a score of at least 80 and above in the Pre-Test for Measuring Head Bath Knowledge Levels, and
* To volunteer to participate in the study.

Exclusion Criteria:

* To not volunteer to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Standardized patient | 3 months
  It is expected that the education method based on standard patient practice will be more effective in change the Spielberger State and Trait Anxiety Scale scores related to head washing skills in nursing students.
  The Spielberger State and Trait Anxiety Inventory is used to collect data about students' anxiety levels. It consists of a total of 40 items and two parts, namely "State Anxiety Inventory" and "Trait Anxiety Inventory". The State and Trait Anxiety Inventory consists of 40 items. The total point value obtained from the scale is between 20-80. A high score indicates a high level of anxiety.
Model with Low Closeness to Reality | 3 months
  It is expected that the Modified Simulation Effectiveness Tool score will be change for the nursing students who practice the skill on the model, whose closeness to reality is low in the teaching of the head bath skill.
  This tool consists of 19 items. The score range of the vehicle is between 18-95. An increase in the score obtained from this tool indicates that the skill performed on the simulation is effective.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University- Faculty of Health Sciences, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cant RP, Cooper SJ. Simulation-based learning in nurse education: systematic review. J Adv Nurs. 2010 Jan;66(1):3-15. doi: 10.1111/j.1365-2648.2009.05240.x. PMID 20423432
- [Background] Alinier G. A typology of educationally focused medical simulation tools. Med Teach. 2007 Oct;29(8):e243-50. doi: 10.1080/01421590701551185. PMID 18236268
- [Background] Bradley P. The history of simulation in medical education and possible future directions. Med Educ. 2006 Mar;40(3):254-62. doi: 10.1111/j.1365-2929.2006.02394.x. PMID 16483328
- [Background] Klipfel JM, Carolan BJ, Brytowski N, Mitchell CA, Gettman MT, Jacobson TM. Patient safety improvement through in situ simulation interdisciplinary team training. Urol Nurs. 2014 Jan-Feb;34(1):39-46. PMID 24716380
- [Background] Leighton K, Ravert P, Mudra V, Macintosh C. Updating the Simulation Effectiveness Tool: Item Modifications and Reevaluation of Psychometric Properties. Nurs Educ Perspect. 2015 Sep-Oct;36(5):317-23. doi: 10.5480/15-1671. PMID 26521501
- [Background] Maran NJ, Glavin RJ. Low- to high-fidelity simulation - a continuum of medical education? Med Educ. 2003 Nov;37 Suppl 1:22-8. doi: 10.1046/j.1365-2923.37.s1.9.x. PMID 14641635
- [Background] McCaughey CS, Traynor MK. The role of simulation in nurse education. Nurse Educ Today. 2010 Nov;30(8):827-32. doi: 10.1016/j.nedt.2010.03.005. Epub 2010 May 16. PMID 20483188
- [Background] Wilford A, Doyle TJ. Integrating simulation training into the nursing curriculum. Br J Nurs. 2006 Sep 28-Oct 11;15(17):926-30. doi: 10.12968/bjon.2006.15.17.21907. PMID 17077785
- [Background] Yoo MS, Yoo IY. The effectiveness of standardized patients as a teaching method for nursing fundamentals. J Nurs Educ. 2003 Oct;42(10):444-8. doi: 10.3928/0148-4834-20031001-06. PMID 14577730
- [Background] Stefanski RR, Rossler KL. Preparing the novice critical care nurse: a community-wide collaboration using the benefits of simulation. J Contin Educ Nurs. 2009 Oct;40(10):443-51; quiz 452-3. doi: 10.3928/00220124-20090923-03. PMID 19831325